CLINICAL TRIAL: NCT03576703
Title: The Influence of Diet During and After Exercise on Metabolic Benefits of Exercise in Overweight Adults
Brief Title: Sugar-sweetened Beverages Influence Benefits of Exercise in Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Principal Investigator, Mary Miles, Professor, Montana State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MW CTR-IN 15-746Q-MSU-PG21-00
Record Dates: First submitted 2018-06-26; First posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Inflammation; Insulin Sensitivity
Keywords: metabolic syndrome; inflammation; insulin sensitivity; metabolic flexibility; overweight/obese
MeSH Terms: conditions — Inflammation; Insulin Resistance; Metabolic Syndrome; Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EX+H2O (Experimental): Exercise and diet that did not include SSB
  Interventions: Other: Exercise with and without SSB ingestion
- EX+SSB (Experimental): Exercise and diet that includes SSB
  Interventions: Other: Exercise with and without SSB ingestion
- CONTROL (No Intervention): No exercise and diet that did not include SSB

INTERVENTIONS:
Other: Exercise with and without SSB ingestion — Consumption of a prescribed diet with and without SSB and performance of moderate aerobic exercise or resting/control
  Arms: EX+H2O; EX+SSB

SUMMARY:
The objective of this study was to determine how metabolic and inflammatory effects of physical exercise in overweight individuals are altered when sugar-sweetened beverages (SSB) are consumed after physical exercise. A randomized, controlled crossover trial was performed in which participants performed exercise with and without the ingestions of SSB during exercise or a non-exercise control condition to evaluate metabolic and inflammatory responses one day after the exercise and or SSB treatment.

DETAILED DESCRIPTION:
Participants: Women (n=24; 18-55 y) with a BMI > 25 and < 35 kg·m-2 who are sedentary to moderately active were recruited to participate. Research Design: This study was a randomized, counter-balanced, cross-over clinical trial consisting of three experimental conditions in which each participant served as her/his own control. Assessments of health history, physical activity (to confirm that participants were physically inactive), anthropometrics, resting metabolic rate, and aerobic capacity were made during an initial laboratory visit. Participants performed three different study conditions, typically separated by one week, thus women were not tested in a specific menstrual cycle phase. Participants recorded their diet the day before and the morning of the first condition and replicated this for the second and third conditions. On the study days, participants consumed their breakfast prior to 9:00 AM and arrived in the lab at 11 AM. The three conditions were performed in randomized order. In the control condition (CON), participants rested quietly for 1 hour. In the remaining two conditions, participants performed 45 minutes of treadmill exercise at 11 AM. Following the rest or exercise period, subjects were provided energy balanced diets. Total energy intake was balanced across exercise conditions and appropriately adjusted for the lack of exercise in the CON condition. At 7 AM on the following morning, following an overnight fast, an oral glucose tolerance test (OGTT) was performed. Measurements were made to determine fasting glucose, insulin and lipid panel, 2-hour OGTT glucose, insulin sensitivity (SI OGTT), early (0-30 min) and late (30-120 min) glucose stimulated insulin secretion (GSIS) based on c-peptide concentrations. Indirect calorimetry was also performed to determine resting carbohydrate and fat oxidation and metabolic flexibility, defined as the change in respiratory exchange ration (RER) during the OGTT. Interleukin-6, tumor necrosis factor-alpha, and reactive oxygen species were measure before, 60, and 120 minutes during the OGTT to assess the inflammation response.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 and < 35 kg/m2
* sedentary to moderately active

Exclusion Criteria:

* inflammatory conditions
* heart disease, diabetes, and other diseases that may interfere with the safety of exercise or other experimental procedures
* allergy to wheat, gluten, dairy, or peanuts
* taking blood pressure, cholesterol lowering, or anti-inflammatory medications
* taking hormone-based birth control with exception of intrauterine device,
* pregnant
* health concerns that make it difficult to participate in study procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2015-07-09 (Actual); Study Completion 2015-07-09 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | 2 hours
  75 g oral glucose tolerance test with measurement of glucose and insulin
Metabolic flexibility | 2 hours
  Change in respiratory exchange ratio in response to ingestion of 75 g of glucose
Inflammation | 2 hours
  Change in cytokine and reactive oxygen species concentrations after ingestion of 75 g of glucose

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Miles, PhD, Principal Investigator — Montana State University

IPD SHARING:
Plan to Share IPD: No